CLINICAL TRIAL: NCT01289262
Title: Long Term Comparison of Double Layer Continuously Locked Closure of Uterine Incision in Cesarean Section Versus Double Layer Purse String Closure (Turan Technique): A Prospective Randomized Study
Brief Title: Long Term Comparison of Two Different Techniques of Uterine Cesarean Incision Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Cem Turan, Chief Clinical, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kartal2; 21.01.2011-02 (02) (Other: Ethics committee ID number)
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section; Complications; Placenta Previa; Placenta Accreta
Keywords: Cesarean section; Kerr incision; Purse string suturing in CS; Continuous locked suturing in CS
MeSH Terms: conditions — Placenta Previa; Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purse string closure technique (Active Comparator): Uterine Kerr incision will be closed with purse string suture.
  Interventions: Procedure: Purse string closure technique
- Continuously locked closure technique (Active Comparator): Uterine Kerr incision will be closed with continuously locked closure technique.
  Interventions: Procedure: Continuously locked closure technique

INTERVENTIONS:
Procedure: Purse string closure technique — Uterine incision will be closed with purse string closure technique.
  Other Names: Uterine incision in C/S
  Arms: Purse string closure technique
Procedure: Continuously locked closure technique — Uterine incision will be closed with continuously locked closure technique
  Other Names: Uterine incision in C/S
  Arms: Continuously locked closure technique

SUMMARY:
Cesarean section (C/S) is an operation most commonly performed in Obstetrics and Gynecology Clinics. Complications related with incomplete healing of Kerr uterine incision after C/S (adhesions, separation (dehiscence), endometritis, endometriosis, anomalous placentation in subsequent pregnancies, incomplete or complete uterine rupture in subsequent pregnancies, ...) are very important issues. Classically Kerr incision is repaired with continuous locked suturing. Purse string suturing of Kerr incision may reduce the size of the incision and in turn may reduce short and long term complications. For this reason, the investigators aimed to compare two closure techniques.

DETAILED DESCRIPTION:
In the clinic, patients undergoing cesarean section that meet the criteria for inclusion into the study and agreed to participate in the study will be randomized into two groups (computer-assisted randomization method will be used.) In the first group of patients classical closure method of Kerr incision(double layered continuously locked suturing) will be used. In the second group of patients double layered purse string closure technique will be used.

Women will be followed for a subsequent pregnancy in the next average 6 years. If they become pregnant again they will be followed up during pregnancy for comparison of long-term effects of the two suture techniques. Patients will be followed especially from the aspects of placental anomalies. Presence of intra-abdominal adhesions, uterine dehiscence, placenta previa, placental invasion anomalies (eg, placenta accreta and others)and incomplete or complete rupture will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term (> 37 weeks) pregnancy
* Cervical dilatation < 4 cm
* Kerr incision
* Age > 18 years old

Exclusion Criteria:

* Being in active phase of labor
* Emergency situations (fetal distress, cord prolapse, placental abruption,severe pre-eclampsia, eclampsia, placenta previa, vasa previa )
* Having a history of uterine surgery (myomectomy, hysterotomy) other than CS
* Extension of Kerr incision
* Multiple pregnancy
* Maternal diabetes mellitus
* Maternal connective tissue disease
* Uterine malformation
* Uterine fibroids on Kerr incision line
* Chorioamnionitis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cem Turan, Study Director — Health Institutes of Turkey ISTANBUL, TURKEY
Locations (1):
- Health Institutes of Turkey ISTANBUL, TURKEY, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Turan C. Long-term follow-up of purse-string double-layer closure (Turan technique) for repairing the uterine incision during cesarean delivery. Am J Obstet Gynecol MFM. 2024 Jan;6(1):101212. doi: 10.1016/j.ajogmf.2023.101212. Epub 2023 Nov 2. No abstract available. PMID 37925053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Started | 84 | 84
Completed | 51 | 65
Not Completed | 33 | 19
Not completed — Lost to Follow-up | 29 | 16
Not completed — Exclusion due to expanded Kerr incision | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique | Total
Number analyzed (Participants) | 51 | 65 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.6 (5.0) | 28.5 (5.3) | 29.05 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 65 | 116
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 51 | 65 | 116

OUTCOME MEASURES:

1. Primary Outcome: Placenta Previa
Description: It will be noted whether placenta previa in cesarean operation of the subsequent pregnancy within next average 6 years, and two groups will be compared.
Time Frame: Subsequent pregnancy within next average 6 years
Population: Eighteen of 51 patients in the study group (purse string) became pregnant. Of the 18 patients in the study group, pregnancy was terminated by cesarean section without low lying placenta, placenta previa marginalis and placenta previa totalis. Of the 65 patients in the control group, 23 became pregnant. Three of them developed low lying placenta, two developed placenta previa marginalis, and one developed placenta previa totalis.
Measure: Count of Participants; unit: Participants
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 18 | 23
Participants
  Subsequent pregnancy without low lying placenta, placenta previa marginalis and totalis | 18 | 17
  Low lying placenta | 0 | 3
  Placenta previa marginalis | 0 | 2
  Placenta previa totalis | 0 | 1

2. Secondary Outcome: Placenta Insertion Anomalies
Description: It will be noted whether placenta insertion anomalies (placenta accreta and others) in cesarean operation of the subsequent pregnancy within next average 6 years, and two groups will be compared.
Time Frame: Subsequent pregnancy within next average 6 years
Population: Placental adhesion (insertion) anomaly did not develop in any of the 18 cases who became pregnant in the Turan technique (purse string) group and in none of the 23 cases who became pregnant in the control (continuously locked closure) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 18 | 23
Participants
  No placental adhesion (insertion) anomaly | 18 | 23
  Placental adhesion (insertion) anomaly | 0 | 0

3. Secondary Outcome: Uterine Rupture
Description: It will be noted whether uterine rupture (incomplete or complete, dehiscence of uterine incision) in cesarean operation of the subsequent pregnancy within next average 6 years, and two groups will be compared.
Time Frame: Subsequent pregnancy within next average 6 years
Population: Uterine rupture (incomplete or complete, dehiscence of uterine incision) did not develop in any of the 18 cases who became pregnant in the Turan technique (Purse string closure technique) group and in none of the 23 cases who became pregnant in the control (continuously locked closure technique) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 18 | 23
Participants
  Without uterine rupture (incomplete or complete, dehiscence of uterine incision) | 18 | 23
  With uterine rupture (incomplete or complete, dehiscence of uterine incision) | 0 | 0

4. Secondary Outcome: Intra-abdominal Adhesions
Description: It will be noted whether intra-abdominal adhesion in cesarean operation of the subsequent pregnancy within next average 6 years, and two groups will be compared.
Time Frame: Up to average 6 years
Population: Intra-abdominal filmy adhesion was detected in 2 of 18 pregnant cases in the Turan technique (purse string) group and intra-abdominal adhesion developed in 6 of 23 cases who became pregnant in the control (Continuously locked closure technique) group. Three of them were filmy and the other three were dense adhesions involving the omentum and intestine.
Measure: Count of Participants; unit: Participants
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
Number analyzed (Participants) | 18 | 23
Participants
  No intra-abdominal adhesions | 16 | 17
  Filmy intra-abdominal adhesions | 2 | 3
  Dense intra-abdominal adhesions | 0 | 3

ADVERSE EVENTS:
Time Frame: 6 years
Description: No Adverse event
Arm/Group | Purse String Closure Technique | Continuously Locked Closure Technique
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/23
Other Adverse Events (participants affected / at risk) | 0/18 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No